CLINICAL TRIAL: NCT01175720
Title: Clinical Comparison Between Two Surgical Techniques With Acellular Dermal Matrix Graft in the Treatment of Gingival Recessions
Brief Title: Clinical Comparison Between Two Surgical Techniques for the Treatment of Gingival Recessions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Arthur Belem Novaes Jr, Clinical comparison between two surgical techniques with acellular dermal matrix graft in the treatment of gingival recessions, University of Sao Paulo
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: lga030183
Record Dates: First submitted 2010-08-03; First posted 2010-08-05 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Gingival Recession
Keywords: gingival recession; acellular dermal matrix graft; root coverage
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- test and control (Experimental): The test and control technique will be tested in a split-mouth design.
  Interventions: Procedure: Periodontal surgery to gingival recessions

INTERVENTIONS:
Procedure: Periodontal surgery to gingival recessions — Test and control technique to treat gingival recessions.

SUMMARY:
The aim of this study is to test a surgical technique for the treatment of gingival recessions. The hypothesis of the study is to promote greater root coverage and better healing.

ELIGIBILITY:
Inclusion Criteria:

* Recession defects are Miller's class I or II and do not vary more or equal than 3 mm
* Main complaint aesthetic issues or dentine hypersensitivity
* The patient must be a candidate for bilateral root coverage procedure
* Patient shows sufficient plaque control (FMPS < 20%)
* The patient is able to comply with the study-related procedures such as exercising good oral hygiene and attending all follow-up procedures
* The patient is able to fully understand the nature of the proposed surgery and is able to provide a signed informed consent

Exclusion Criteria:

* Smokers
* Systemic diseases
* Pregnants or lactating
* Periodontal disease
* General contraindications for dental and/or surgical treatment are present
* The patient has a history of malignancy, radiotherapy, or chemotherapy for malignancy within the past five years
* The patient is taking medications or having treatments which have an effect on mucosal healing in general (e.g. steroids, large doses of anti-inflammatory drugs)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-08; Primary Completion 2011-06 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Percentage of root coverage | 6 months
  Clinical parameters will be assessed after 6 months of surgical procedures.

SECONDARY OUTCOMES:
Keratinized Tissue | 6 months
  Clinical parameters will be assessed after 6 months of surgical procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Arthur B. Novaes Júnior, PhD, Principal Investigator — University of Sao Paulo; Lauro G. Ayub, MSD student, Principal Investigator — University of Sao Paulo
Locations (1):
- Faculty of Dentistry of Ribeirão Preto USP, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Derived] Ayub LG, Ramos UD, Reino DM, Grisi MF, Taba M Jr, Souza SL, Palioto DB, Novaes AB Jr. A Randomized comparative clinical study of two surgical procedures to improve root coverage with the acellular dermal matrix graft. J Clin Periodontol. 2012 Sep;39(9):871-8. doi: 10.1111/j.1600-051X.2012.01915.x. Epub 2012 Jun 19. PMID 22712624